CLINICAL TRIAL: NCT00902720
Title: Ovarian Tissue Freezing For Fertility Preservation In Women Facing A Fertility Threatening Medical Diagnosis Or Treatment Regimen: A Study By The National Physicians Cooperative of the Oncofertility Consortium At Northwestern University
Brief Title: Ovarian Tissue Freezing For Fertility Preservation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David M Lee, MD, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: U54RR024347; U54RR024347 (Other Grant/Funding Number: NIH); IRB00005031 (Other: OHSU)
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Malignancy; Fertility
Keywords: Ovarian; Tissue; Cryopreservation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cryopreservation (Experimental): The ovarian tissue is frozen and banked at the in vitro fertilization lab at the Center for Health and Healing at OHSU.
  Interventions: Other: Tissue sample storage

INTERVENTIONS:
Other: Tissue sample storage — The tissue sample is frozen and held at -140 degrees at the in vitro fertilization lab at the Center for Health and Healing at OHSU.

SUMMARY:
The purpose of this study is to offer an alternative method to women who wish to preserve the possibility of fertility, as well as to learn more about the ability of human eggs to survive and function after long term storage in frozen ovaries (ovarian tissue cryopreservation). The study will seek to preserve ovarian tissue and reproductive potential for patients whose medical or surgical treatment may harm ovaries or remove ovarian tissue.

DETAILED DESCRIPTION:
Women who have not yet undergone this procedure, and who present to the Fertility Consultants desiring fertility preservation, will be offered participation in the study.

Subjects will undergo an initial visit which will include a blood draw, ultrasound, and any additional tests or exams that are medically indicated for the subject's diagnosis in preparation for surgery. Subjects will then undergo an oophorectomy surgery (removal of one or both ovaries). Following removal, subject's ovarian tissue will be cryopreserved (frozen) and stored for possible future use. We also plan to collect subjects medical history information to enter into a research database. Subjects will be followed until they decide to use their tissue for fertility purposes.

We will also retrospectively enroll women who have already undergone this procedure by contacting them by mail and offering participation in our ovarian tissue cryopreservation database.

ELIGIBILITY:
Inclusion Criteria:

* Woman between the age of 18-41 years who will undergo surgery, chemotherapy, drug treatment and/or radiation for the treatment or prevention of a medical condition or malignancy expected to result in permanent and complete loss of subsequent ovarian function or have a medical condition or malignancy that requires removal of all or part of one or both ovaries.
* Patients may have newly diagnosed or recurrent disease. Those who were not enrolled at the time of initial diagnosis are eligible if they have not received therapy that is viewed as likely to result in complete and permanent loss of ovarian function.
* For patients undergoing elective removal of an ovary for fertility preservation only, have two ovaries.
* Patients who already have stored cryopreserved ovarian tissue in a frozen state prior to undergoing cancer treatments (surgery, chemotherapy or radiation) will be eligible for enrollment with informed consent.
* Signed an approved informed consent and authorization permitting the release of personal health information. The patient and/or the patient's legally authorized guardian must acknowledge in writing that consent for specimen collection has been obtained, in accordance with institutional policies approved by the U.S. Department of Health and Human Services.

Exclusion Criteria:

* Women with psychological, psychiatric, or other conditions which prevent giving fully informed consent.
* Women whose underlying medical condition significantly increases their risk of complications from anesthesia and surgery.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
This study will provide a pool of research ovarian tissue to use to develop and test methods to expand the range of fertility preservation options available to female cancer patients. | May 2009 - January 2010

SECONDARY OUTCOMES:
Optimize techniques for freezing and thawing of ovarian tissue for use in transplant or in vitro follicle maturation (IFM). | May 2009 - January 2010
Investigate factors affecting successful maturation of immature follicles obtained from ovarian tissue including the use of 3-dimensional biogel scaffolds, growth factors, hormones and other culture conditions. | May 2009 - January 2010
Determine the efficacy of ovarian cryopreservation techniques. | May 2009 - January 2010
Provide long term follow up on patients who have ovarian tissue frozen for their own use. | May 2009 - January 2010
A substantial portion of the patient's tissue will be cryopreserved and reserved for her own use. | May 2009 - January 2010

CONTACTS AND LOCATIONS:
Overall Officials: David M Lee, MD, Principal Investigator — Oregon Health and Sciences University
Locations (1):
- Oregon Health and Sciences Universtiy, Portland, Oregon, United States

REFERENCES:
- [Background] Blatt J. Pregnancy outcome in long-term survivors of childhood cancer. Med Pediatr Oncol. 1999 Jul;33(1):29-33. doi: 10.1002/(sici)1096-911x(199907)33:13.0.co;2-2. PMID 10401494
- [Background] Meirow D, Nugent D. The effects of radiotherapy and chemotherapy on female reproduction. Hum Reprod Update. 2001 Nov-Dec;7(6):535-43. doi: 10.1093/humupd/7.6.535. PMID 11727861
- [Background] Greenlee RT, Murray T, Bolden S, Wingo PA. Cancer statistics, 2000. CA Cancer J Clin. 2000 Jan-Feb;50(1):7-33. doi: 10.3322/canjclin.50.1.7. PMID 10735013
- [Background] Meirow D. Ovarian injury and modern options to preserve fertility in female cancer patients treated with high dose radio-chemotherapy for hemato-oncological neoplasias and other cancers. Leuk Lymphoma. 1999 Mar;33(1-2):65-76. doi: 10.3109/10428199909093726. PMID 10194122
- [Background] Meirow D. Epidemiology and infertility in cancer patients. In: Gosden R, Tulandi T, editors. Preservation of fertility. London: Taylor and Francis, 2004:21-38.
- [Background] Koyama H, Wada T, Nishizawa Y, Iwanaga T, Aoki Y. Cyclophosphamide-induced ovarian failure and its therapeutic significance in patients with breast cancer. Cancer. 1977 Apr;39(4):1403-9. doi: 10.1002/1097-0142(197704)39:43.0.co;2-8. PMID 851940
- [Background] Goldhirsch A, Gelber RD, Castiglione M. The magnitude of endocrine effects of adjuvant chemotherapy for premenopausal breast cancer patients. The International Breast Cancer Study Group. Ann Oncol. 1990;1(3):183-8. doi: 10.1093/oxfordjournals.annonc.a057718. PMID 2261364
- [Background] Chiarelli AM, Marrett LD, Darlington G. Early menopause and infertility in females after treatment for childhood cancer diagnosed in 1964-1988 in Ontario, Canada. Am J Epidemiol. 1999 Aug 1;150(3):245-54. doi: 10.1093/oxfordjournals.aje.a009995. PMID 10430228
- [Background] Falcone T, Attaran M, Bedaiwy MA, Goldberg JM. Ovarian function preservation in the cancer patient. Fertil Steril. 2004 Feb;81(2):243-57. doi: 10.1016/j.fertnstert.2003.06.031. PMID 14967351
- [Background] Wallace WH, Thomson AB, Saran F, Kelsey TW. Predicting age of ovarian failure after radiation to a field that includes the ovaries. Int J Radiat Oncol Biol Phys. 2005 Jul 1;62(3):738-44. doi: 10.1016/j.ijrobp.2004.11.038. PMID 15936554
- [Background] Critchley HO, Wallace WH, Shalet SM, Mamtora H, Higginson J, Anderson DC. Abdominal irradiation in childhood; the potential for pregnancy. Br J Obstet Gynaecol. 1992 May;99(5):392-4. doi: 10.1111/j.1471-0528.1992.tb13755.x. PMID 1622911
- [Background] Bath LE, Critchley HO, Chambers SE, Anderson RA, Kelnar CJ, Wallace WH. Ovarian and uterine characteristics after total body irradiation in childhood and adolescence: response to sex steroid replacement. Br J Obstet Gynaecol. 1999 Dec;106(12):1265-72. doi: 10.1111/j.1471-0528.1999.tb08180.x. PMID 10609720
- [Background] Rappaport R, Brauner R, Czernichow P, Thibaud E, Renier D, Zucker JM, Lemerle J. Effect of hypothalamic and pituitary irradiation on pubertal development in children with cranial tumors. J Clin Endocrinol Metab. 1982 Jun;54(6):1164-8. doi: 10.1210/jcem-54-6-1164. PMID 6804477
- [Background] Davies HA, Didcock E, Didi M, Ogilvy-Stuart A, Wales JK, Shalet SM. Growth, puberty and obesity after treatment for leukaemia. Acta Paediatr Suppl. 1995 Sep;411:45-50; discussion 51. doi: 10.1111/j.1651-2227.1995.tb13862.x. PMID 8563069
- [Background] Ogilvy-Stuart AL, Clayton PE, Shalet SM. Cranial irradiation and early puberty. J Clin Endocrinol Metab. 1994 Jun;78(6):1282-6. doi: 10.1210/jcem.78.6.8200926.
- [Background] Kwon JS, Case AM. Preserving reproductive function in women with cancer. Sexuality,Reproduction & Menopause 2004;2(2):222-229. (A Publication of the American Society for Reproductive Medicine) http://www.srmjournal.org/home
- [Background] Blumenfeld Z. Preservation of fertility and ovarian function and minimalization of chemotherapy associated gonadotoxicity and premature ovarian failure: the role of inhibin-A and -B as markers. Mol Cell Endocrinol. 2002 Feb 22;187(1-2):93-105. doi: 10.1016/s0303-7207(01)00712-2. PMID 11988316
- [Background] Revel A, Laufer N. Protecting female fertility from cancer therapy. Mol Cell Endocrinol. 2002 Feb 22;187(1-2):83-91. doi: 10.1016/s0303-7207(01)00705-5. PMID 11988315
- [Background] Ataya K, Pydyn E, Ramahi-Ataya A, Orton CG. Is radiation-induced ovarian failure in rhesus monkeys preventable by luteinizing hormone-releasing hormone agonists?: Preliminary observations. J Clin Endocrinol Metab. 1995 Mar;80(3):790-5. doi: 10.1210/jcem.80.3.7883832.
- [Background] Ataya K, Rao LV, Lawrence E, Kimmel R. Luteinizing hormone-releasing hormone agonist inhibits cyclophosphamide-induced ovarian follicular depletion in rhesus monkeys. Biol Reprod. 1995 Feb;52(2):365-72. doi: 10.1095/biolreprod52.2.365. PMID 7711205
- [Background] Blumenfeld Z, Avivi I, Linn S, Epelbaum R, Ben-Shahar M, Haim N. Prevention of irreversible chemotherapy-induced ovarian damage in young women with lymphoma by a gonadotrophin-releasing hormone agonist in parallel to chemotherapy. Hum Reprod. 1996 Aug;11(8):1620-6. doi: 10.1093/oxfordjournals.humrep.a019457. PMID 8921104
- [Background] Waxman JH, Ahmed R, Smith D, Wrigley PF, Gregory W, Shalet S, Crowther D, Rees LH, Besser GM, Malpas JS, et al. Failure to preserve fertility in patients with Hodgkin's disease. Cancer Chemother Pharmacol. 1987;19(2):159-62. doi: 10.1007/BF00254570. PMID 3105906
- [Background] Oktay K, Cil AP, Bang H. Efficiency of oocyte cryopreservation: a meta-analysis. Fertil Steril. 2006 Jul;86(1):70-80. doi: 10.1016/j.fertnstert.2006.03.017. PMID 16818031
- [Background] Porcu E, Fabbri R, Damiano G, Giunchi S, Fratto R, Ciotti PM, Venturoli S, Flamigni C. Clinical experience and applications of oocyte cryopreservation. Mol Cell Endocrinol. 2000 Nov 27;169(1-2):33-7. doi: 10.1016/s0303-7207(00)00348-8. PMID 11155951
- [Background] Fabbri R, Porcu E, Marsella T, Rocchetta G, Venturoli S, Flamigni C. Human oocyte cryopreservation: new perspectives regarding oocyte survival. Hum Reprod. 2001 Mar;16(3):411-6. doi: 10.1093/humrep/16.3.411. PMID 11228204
- [Background] Borini A, Bonu MA, Coticchio G, Bianchi V, Cattoli M, Flamigni C. Pregnancies and births after oocyte cryopreservation. Fertil Steril. 2004 Sep;82(3):601-5. doi: 10.1016/j.fertnstert.2004.04.025. PMID 15374702
- [Background] Eppig JJ, O'Brien MJ. Development in vitro of mouse oocytes from primordial follicles. Biol Reprod. 1996 Jan;54(1):197-207. doi: 10.1095/biolreprod54.1.197. PMID 8838017
- [Background] Cha KY, Chung HM, Lim JM, Ko JJ, Han SY, Choi DH, Yoon TK. Freezing immature oocytes. Mol Cell Endocrinol. 2000 Nov 27;169(1-2):43-7. doi: 10.1016/s0303-7207(00)00350-6. PMID 11155953
- [Background] Parrott JA, Skinner MK. Direct actions of kit-ligand on theca cell growth and differentiation during follicle development. Endocrinology. 1997 Sep;138(9):3819-27. doi: 10.1210/endo.138.9.5368. PMID 9275070
- [Background] Elvin JA, Yan C, Wang P, Nishimori K, Matzuk MM. Molecular characterization of the follicle defects in the growth differentiation factor 9-deficient ovary. Mol Endocrinol. 1999 Jun;13(6):1018-34. doi: 10.1210/mend.13.6.0309. PMID 10379899
- [Background] Nilsson E, Parrott JA, Skinner MK. Basic fibroblast growth factor induces primordial follicle development and initiates folliculogenesis. Mol Cell Endocrinol. 2001 Apr 25;175(1-2):123-30. doi: 10.1016/s0303-7207(01)00391-4. PMID 11325522
- [Background] Otsuka F, Moore RK, Shimasaki S. Biological function and cellular mechanism of bone morphogenetic protein-6 in the ovary. J Biol Chem. 2001 Aug 31;276(35):32889-95. doi: 10.1074/jbc.M103212200. Epub 2001 Jul 10. PMID 11447221
- [Background] Nilsson EE, Kezele P, Skinner MK. Leukemia inhibitory factor (LIF) promotes the primordial to primary follicle transition in rat ovaries. Mol Cell Endocrinol. 2002 Feb 25;188(1-2):65-73. doi: 10.1016/s0303-7207(01)00746-8. PMID 11911947
- [Background] Yoon SJ, Kim KH, Chung HM, Choi DH, Lee WS, Cha KY, Lee KA. Gene expression profiling of early follicular development in primordial, primary, and secondary follicles. Fertil Steril. 2006 Jan;85(1):193-203. doi: 10.1016/j.fertnstert.2005.07.1296. PMID 16412753
- [Background] Gougeon A. Regulation of ovarian follicular development in primates: facts and hypotheses. Endocr Rev. 1996 Apr;17(2):121-55. doi: 10.1210/edrv-17-2-121. No abstract available. PMID 8706629
- [Background] Zeleznik AJ. The physiology of follicle selection. Reprod Biol Endocrinol. 2004 Jun 16;2:31. doi: 10.1186/1477-7827-2-31. PMID 15200680
- [Background] Kreeger PK, Fernandes NN, Woodruff TK, Shea LD. Regulation of mouse follicle development by follicle-stimulating hormone in a three-dimensional in vitro culture system is dependent on follicle stage and dose. Biol Reprod. 2005 Nov;73(5):942-50. doi: 10.1095/biolreprod.105.042390. Epub 2005 Jun 29. PMID 15987824
- [Background] Kreeger PK, Deck JW, Woodruff TK, Shea LD. The in vitro regulation of ovarian follicle development using alginate-extracellular matrix gels. Biomaterials. 2006 Feb;27(5):714-23. doi: 10.1016/j.biomaterials.2005.06.016. Epub 2005 Aug 1. PMID 16076485
- [Background] Pangas SA, Saudye H, Shea LD, Woodruff TK. Novel approach for the three-dimensional culture of granulosa cell-oocyte complexes. Tissue Eng. 2003 Oct;9(5):1013-21. doi: 10.1089/107632703322495655. PMID 14633385
- [Background] Xu M, West E, Shea LD, Woodruff TK. Identification of a stage-specific permissive in vitro culture environment for follicle growth and oocyte development. Biol Reprod. 2006 Dec;75(6):916-23. doi: 10.1095/biolreprod.106.054833. Epub 2006 Sep 6. PMID 16957022
- [Background] Xu M, Kreeger PK, Shea LD, Woodruff TK. Tissue-engineered follicles produce live, fertile offspring. Tissue Eng. 2006 Oct;12(10):2739-46. doi: 10.1089/ten.2006.12.2739. PMID 17518643
- [Background] Oktay K, Nugent D, Newton H, Salha O, Chatterjee P, Gosden RG. Isolation and characterization of primordial follicles from fresh and cryopreserved human ovarian tissue. Fertil Steril. 1997 Mar;67(3):481-6. doi: 10.1016/s0015-0282(97)80073-8. PMID 9091334
- [Background] Gosden RG, Baird DT, Wade JC, Webb R. Restoration of fertility to oophorectomized sheep by ovarian autografts stored at -196 degrees C. Hum Reprod. 1994 Apr;9(4):597-603. doi: 10.1093/oxfordjournals.humrep.a138556. PMID 8046009
- [Background] Yeoman RR, Wolf DP, Lee DM. Coculture of monkey ovarian tissue increases survival after vitrification and slow-rate freezing. Fertil Steril. 2005 Apr;83 Suppl 1:1248-54. doi: 10.1016/j.fertnstert.2004.11.036. PMID 15831299
- [Background] DEANESLY R. Immature rat ovaries grafted after freezing and thawing. J Endocrinol. 1954 Aug;11(2):197-200. doi: 10.1677/joe.0.0110197. No abstract available. PMID 13201707
- [Background] PARKES AS, SMITH AU. Preservation of ovarian tissue at -79 degrees C. for transplantation. Acta Endocrinol (Copenh). 1954;17(1-4):313-20. No abstract available. PMID 13227843
- [Background] MUSSETT MV, PARROTT DM. Factors affecting the fertility of mice with orthotopic ovarian grafts. J Reprod Fertil. 1961 Feb;2:80-97. doi: 10.1530/jrf.0.0020080. No abstract available. PMID 13727124
- [Background] Oktay K, Aydin BA, Karlikaya G. A technique for laparoscopic transplantation of frozen-banked ovarian tissue. Fertil Steril. 2001 Jun;75(6):1212-6. doi: 10.1016/s0015-0282(01)01776-9. PMID 11384651
- [Background] Donnez J, Dolmans MM, Demylle D, Jadoul P, Pirard C, Squifflet J, Martinez-Madrid B, van Langendonckt A. Livebirth after orthotopic transplantation of cryopreserved ovarian tissue. Lancet. 2004 Oct 16-22;364(9443):1405-10. doi: 10.1016/S0140-6736(04)17222-X. PMID 15488215
- [Background] Silber SJ, Lenahan KM, Levine DJ, Pineda JA, Gorman KS, Friez MJ, Crawford EC, Gosden RG. Ovarian transplantation between monozygotic twins discordant for premature ovarian failure. N Engl J Med. 2005 Jul 7;353(1):58-63. doi: 10.1056/NEJMoa043157. Epub 2005 Jun 7. PMID 15941849
- [Background] Oktay K, Economos K, Kan M, Rucinski J, Veeck L, Rosenwaks Z. Endocrine function and oocyte retrieval after autologous transplantation of ovarian cortical strips to the forearm. JAMA. 2001 Sep 26;286(12):1490-3. doi: 10.1001/jama.286.12.1490. PMID 11572742
- [Background] Lee DM, Yeoman RR, Battaglia DE, Stouffer RL, Zelinski-Wooten MB, Fanton JW, Wolf DP. Live birth after ovarian tissue transplant. Nature. 2004 Mar 11;428(6979):137-8. doi: 10.1038/428137a. PMID 15014485
- [Background] Harp R, Leibach J, Black J, Keldahl C, Karow A. Cryopreservation of murine ovarian tissue. Cryobiology. 1994 Aug;31(4):336-43. doi: 10.1006/cryo.1994.1040. PMID 7924392
- [Background] Sztein J, Sweet H, Farley J, Mobraaten L. Cryopreservation and orthotopic transplantation of mouse ovaries: new approach in gamete banking. Biol Reprod. 1998 Apr;58(4):1071-4. doi: 10.1095/biolreprod58.4.1071. PMID 9546742
- [Background] Schnorr JA OS, Toner JP, Hsiu JG, Willams RF, Hodgen GD. Fresh and cryopreserved extrapelvic ovarian transplantation in non-human primates: folliculogenesis, ovulation, corpus luteum function, endometrial development, and menstrual patterns. Abstract presented at: the American Society of Reproductive Medicine 2000 Annual Meeting; October 21-26, 2000; San Diego, California
- [Background] Gougeon A, Ecochard R, Thalabard JC. Age-related changes of the population of human ovarian follicles: increase in the disappearance rate of non-growing and early-growing follicles in aging women. Biol Reprod. 1994 Mar;50(3):653-63. doi: 10.1095/biolreprod50.3.653. PMID 8167237
- [Background] Gougeon A. Ovarian follicular growth in humans: ovarian ageing and population of growing follicles. Maturitas. 1998 Oct 12;30(2):137-42. doi: 10.1016/s0378-5122(98)00069-3. PMID 9871908
- [Background] Oktay K, Karlikaya G. Ovarian function after transplantation of frozen, banked autologous ovarian tissue. N Engl J Med. 2000 Jun 22;342(25):1919. doi: 10.1056/NEJM200006223422516. No abstract available. PMID 10877641
- [Background] Radford JA, Lieberman BA, Brison DR, Smith AR, Critchlow JD, Russell SA, Watson AJ, Clayton JA, Harris M, Gosden RG, Shalet SM. Orthotopic reimplantation of cryopreserved ovarian cortical strips after high-dose chemotherapy for Hodgkin's lymphoma. Lancet. 2001 Apr 14;357(9263):1172-5. doi: 10.1016/s0140-6736(00)04335-x. PMID 11323045
- [Background] Oktay K, Buyuk E, Veeck L, Zaninovic N, Xu K, Takeuchi T, Opsahl M, Rosenwaks Z. Embryo development after heterotopic transplantation of cryopreserved ovarian tissue. Lancet. 2004 Mar 13;363(9412):837-40. doi: 10.1016/S0140-6736(04)15728-0. PMID 15031026
- [Background] Meirow D, Levron J, Eldar-Geva T, Hardan I, Fridman E, Zalel Y, Schiff E, Dor J. Pregnancy after transplantation of cryopreserved ovarian tissue in a patient with ovarian failure after chemotherapy. N Engl J Med. 2005 Jul 21;353(3):318-21. doi: 10.1056/NEJMc055237. Epub 2005 Jun 27. No abstract available. PMID 15983020
- [Background] Demeestere I, Simon P, Buxant F, Robin V, Fernandez SA, Centner J, Delbaere A, Englert Y. Ovarian function and spontaneous pregnancy after combined heterotopic and orthotopic cryopreserved ovarian tissue transplantation in a patient previously treated with bone marrow transplantation: case report. Hum Reprod. 2006 Aug;21(8):2010-4. doi: 10.1093/humrep/del092. Epub 2006 Apr 3. PMID 16585122
- [Background] Leporrier M, von Theobald P, Roffe JL, Muller G. A new technique to protect ovarian function before pelvic irradiation. Heterotopic ovarian autotransplantation. Cancer. 1987 Nov 1;60(9):2201-4. doi: 10.1002/1097-0142(19871101)60:93.0.co;2-z. PMID 3440230
- [Background] Wang X, Chen H, Yin H, Kim SS, Lin Tan S, Gosden RG. Fertility after intact ovary transplantation. Nature. 2002 Jan 24;415(6870):385. doi: 10.1038/415385a. PMID 11807540
- [Background] Bedaiwy MA, Jeremias E, Gurunluoglu R, Hussein MR, Siemianow M, Biscotti C, Falcone T. Restoration of ovarian function after autotransplantation of intact frozen-thawed sheep ovaries with microvascular anastomosis. Fertil Steril. 2003 Mar;79(3):594-602. doi: 10.1016/s0015-0282(02)04842-2. PMID 12620446
- [Background] Imhof M, Bergmeister H, Lipovac M, Rudas M, Hofstetter G, Huber J. Orthotopic microvascular reanastomosis of whole cryopreserved ovine ovaries resulting in pregnancy and live birth. Fertil Steril. 2006 Apr;85 Suppl 1:1208-15. doi: 10.1016/j.fertnstert.2005.11.030. PMID 16616094
- [Background] Shaw JM, Bowles J, Koopman P, Wood EC, Trounson AO. Fresh and cryopreserved ovarian tissue samples from donors with lymphoma transmit the cancer to graft recipients. Hum Reprod. 1996 Aug;11(8):1668-73. doi: 10.1093/oxfordjournals.humrep.a019467. PMID 8921114
- [Background] Kim SS, Hwang IT, Lee HC. Heterotopic autotransplantation of cryobanked human ovarian tissue as a strategy to restore ovarian function. Fertil Steril. 2004 Oct;82(4):930-2. doi: 10.1016/j.fertnstert.2004.02.137. PMID 15482772
- [Background] Sonmezer M, Shamonki MI, Oktay K. Ovarian tissue cryopreservation: benefits and risks. Cell Tissue Res. 2005 Oct;322(1):125-32. doi: 10.1007/s00441-005-1098-4. Epub 2005 Nov 3. PMID 15912406
- [Background] Lee DM, Yeoman RR, Yu T, et al. Sphingosine-1-phosphate inhibits apoptosis in rhesus monkey ovarian tissue in vitro and may improve reproductive function in xenografts. 2005 Joint American Society for Reproductive Medicine/Canadian Fertility & Andrology Society Meeting, Oct. 15-19, Montreal, Quebec, CANADA. Fertil Steril 2005;84(Suppl 1):S2
- [Background] Gunasena KT, Lakey JR, Villines PM, Critser ES, Critser JK. Allogeneic and xenogeneic transplantation of cryopreserved ovarian tissue to athymic mice. Biol Reprod. 1997 Aug;57(2):226-31. doi: 10.1095/biolreprod57.2.226. PMID 9241035
- [Background] Snow M, Cox SL, Jenkin G, Trounson A, Shaw J. Generation of live young from xenografted mouse ovaries. Science. 2002 Sep 27;297(5590):2227. doi: 10.1126/science.1073693. No abstract available. PMID 12351780
- [Background] Weissman A, Gotlieb L, Colgan T, Jurisicova A, Greenblatt EM, Casper RF. Preliminary experience with subcutaneous human ovarian cortex transplantation in the NOD-SCID mouse. Biol Reprod. 1999 Jun;60(6):1462-7. doi: 10.1095/biolreprod60.6.1462. PMID 10330106
- [Background] Kim SS, Soules M, Gosden RG, et al. The evidence of follicle maturation and subsequent ovulation in human ovarian tissue xenografted into severe combined immunodeficient (SCID)mice. Fertil Steril 2000;74:S34
- [Background] Nisolle M, Casanas-Roux F, Qu J, Motta P, Donnez J. Histologic and ultrastructural evaluation of fresh and frozen-thawed human ovarian xenografts in nude mice. Fertil Steril. 2000 Jul;74(1):122-9. doi: 10.1016/s0015-0282(00)00548-3. PMID 10899508
- [Background] Oktay K, Newton H, Gosden RG. Transplantation of cryopreserved human ovarian tissue results in follicle growth initiation in SCID mice. Fertil Steril. 2000 Mar;73(3):599-603. doi: 10.1016/s0015-0282(99)00548-8. PMID 10689020
- [Background] Lee K, Lee S, SJ Y, et al. Resumption of the human primordial follicle growth in xenografts after vitrification of the ovarian tissues. Fertil Steril 2000;74(3 Suppl 1):S214
- [Background] Kim SS, Kang HG, Kim NH, Lee HC, Lee HH. Assessment of the integrity of human oocytes retrieved from cryopreserved ovarian tissue after xenotransplantation. Hum Reprod. 2005 Sep;20(9):2502-8. doi: 10.1093/humrep/dei099. Epub 2005 Jun 9. PMID 15946997
- See also: Related Info — http://www.ohsuwomenshealth.com/research/index.html